CLINICAL TRIAL: NCT05306210
Title: Forxiga Tablets 5mg, 10mgGeneral Drug Use-Results Study n in Chronic Kidney Disease (CKD) Patients
Brief Title: Forxiga CKD Japan Post-Marketing Surveillance (PMS)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D169AC00007
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To capture safety when Forxige is administrated to CKD patients in the real world setting

DETAILED DESCRIPTION:
The purpose of the study is to review the following points during use of Forxiga Tablets (hereinafter referred to as Forxiga) in the real world setting after launch for treatment of CKD.

1. ADRs which are unexpected from the precautions for use in our JPI
2. Understanding of incidence of ADRs during use of Forxiga in the real world setting
3. Factors (ie demography, treatment) possibly having an impact on the safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD except for dialysis and/or renal failure chronic

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who initiate Forxiga treatment for chronic kidney disease aligned with the approved Japanese label for the first time
Sampling Method: Non-Probability Sample
Enrollment: 1029 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence of ADRs during use of Forxiga in the real world setting | from baseline of 1year
  To be calculated incidence of ADRs related to Forxiga during the observation period
Incidence of ADRs which are unexpected from the precautions for use in our JPI | from baseline to 1 year
  To be calculated incidence of ADRs related to Forxiga during the observation period not expected from the precautions for use of Forxiga JPI
Factors (ie demography, treatment) possibly having an impact on the safety | from baseline to 1 year
  Factors which may impact incidence of ADRs analysed by patient demographic characteristic (past medical history and concomitant disease etc)

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — Astrazeneca KK
Locations (46):
- Japan (46):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before a accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169AC00007&attachmentIdentifier=7bd07808-fc52-489d-abb9-5d86e3c3c1a9&fileName=D169AC00007_Redacted_CSR_Synopsis.pdf&versionIdentifier=